CLINICAL TRIAL: NCT05401201
Title: Dual-light Antibacterial Photodynamic Therapy as an Adjunctive Treatment to Topical Corticosteroid Treatment in Patients With Gingival Involvement of Oral Lichen Planus - a Randomized Study
Brief Title: Dual-light Antibacterial Photodynamic Therapy as an Adjunctive Treatment to Corticosteroid Treatment in OLP
Acronym: RELIEF-OLP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koite Health Oy (Industry)
Collaborators: Wellbeing Services County of Pirkanmaa (Other); Tampere University (Other); University of Helsinki (Other); Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OLP-01TRE
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Oral Lichen Planus; Dental Plaque; Oral Bacterial Infection
Keywords: Lumoral; Lumorinse; Plaque; Oral Lichen Planus; aMMP-8; aPDT; Pain score (VAS)
MeSH Terms: conditions — Lichen Planus, Oral; Dental Plaque; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: A total of 60 subjects with histologically confirmed diagnosis of OLP with gingival involvement are enrolled to the study. The subjects are randomized to a study group and a control group. Both groups will use topical corticosteroid treatment for two weeks. In addition, the study group will use Lumoral-device initially once a day.
Masking Description: A sealed envelope system shall be used for randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Subjects in the study group will use the Lumoral device five to seven times a week according to the verbal and written instructions provided to them. In addition, they will brush their teeth twice daily in their customary manner while using the provided sonic toothbrush and regular toothpaste.
  Interventions: Device: Lumoral treatment; Other: Standard oral hygiene self care
- Control group (Active Comparator): Subjects in the control group will brush their teeth in their customary manner twice daily while using the provided sonic toothbrush and regular toothpaste. They will not receive any additional intervention.
  Interventions: Other: Standard oral hygiene self care

INTERVENTIONS:
Device: Lumoral treatment — The investigational Lumoral treatment -device provides a constant and repeatable application which can be done at home and is easily available. All subjects in the study group will receive their own Lumoral treatment -device and Lumorinse-mouth rinse tablets for the complete duration of the study.
  Other Names: Lumorinse mouth rinse
  Arms: Study group
Other: Standard oral hygiene self care — Both groups shall be given oral and written instructions for twice-daily standard oral hygiene self care.
  Other Names: Sonic toothbrush provided

SUMMARY:
This study is designed to investigate the effectiveness of plaque control intervention by home-use dual-light aPDT Lumoral -device as an adjunctive or alternative treatment to triamcinolone acetonide (TCA) mouth rinse or other topical corticosteroid treatment on the symptoms and clinical appearance of symptomatic gingival involvement of oral lichen planus (OLP).

DETAILED DESCRIPTION:
Oral Lichen Planus (OLP) is a relatively common, chronic immune-mediated mucocutaneous disease,that usually occurs on the oral mucosa surfaces. Oral lesions are commonly multiple with a bilateral and symmetrical localization. Most affected sites in the oral cavity are the buccal and lingual mucosa, and the gingiva. Approximately 10% of patients with OLP present manifestations in the gingiva.

Lumoral is a CE-marked medical device developed to provide a potent, targeted antibacterial action on dental plaque in a home environment. The device mechanism of action is antibacterial photodynamic therapy (aPDT). The device is used by swishing a mouth rinse, which has a strong adherence to dental plaque. The plaque-adhered photoactive mouth rinse can be activated by a simple to use light applicator. Use of the device can improve supragingival plaque control. Preliminary results have shown a promising anti-inflammatory response in addition to plaque reduction.

A total of 60 subjects with histologically confirmed diagnosis of OLP with gingival involvement are enrolled to the study. The subjects are randomized to a study group and a control group. Both groups will use topical corticosteroid treatment for two weeks. In addition, the study group will use Lumoral-device initially once a day.

All the subjects shall be assessed for desquamative gingivitis clinical score (DGCS), Escudier Index (EI), visible plaque index (VPI), bleeding on probing index (BOP), pain score (VAS), aMMP-8 inflammation marker and oral candidosis. These analyses shall be performed at baseline and at 4 week, 3, 6 and 12 months after the treatment started.

In addition, psychosocial factors shall be assessed by the graded chronic pain scale (GCPS), the oral health impact profile (OHIP-14) and the generalized anxiety disorder (GAD-7) questionnaires at baseline and at 6 and 12 months after the treatment initiation.

Primary outcome is improvement in average Pain score (VAS) symptom diary during the 12 month study period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of OLP with bilateral symmetrical lesions and gingival involvement
* Able to provide a written consent
* Willing and able to complete questionnaires
* Able to co-operate with the treatment protocol and avoid any other oral hygiene measures outside of the study protocol

Exclusion Criteria:

* Lichenoid lesions suspected to be induced by contact allergy or drugs
* Any treatment for OLP in two weeks prior to the study/ a history of topical therapy for OLP in the past 2 weeks or systemic therapy in the past 4 weeks;
* Pregnant or lactating
* Photosensitivity
* Use of antibiotics within 2 weeks prior the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain score symptom diary (based on Visual Analogue Scale - VAS) | 12 months
  Improvement in average Pain score (VAS) symptom diary during the 12 month study period.
  Assessments:
  1. '365 Average pain score' (VAS) is determined by calculating the average of the pain scores marked in the diary during the total surveillance period of one year;
  2. '52 Average pain score' (VAS) is determined by calculating the average of the pain scores of calendar weeks during the total surveillance period of one year;
  3. 'Positive 52 Average pain score' (VAS) is determined by including the '52 Average pain scores' of those calendar weeks, which have VAS average over 2.

SECONDARY OUTCOMES:
aMMP-8 | 12 Months
  Reduction in inflammation marker aMMP-8 measured by Periosafe®
Visible plaque index (VPI) | 12 Months
  Improvement in visible plaque index (VPI)
Bleeding on probing index (BOP) | 12 Months
  Improvement in the bleeding on probing index (BOP)
Escudier Index (EI) | 12 Months
  Improvement in OLP measured by the Escudier Index (EI)
Visual Analogue Scale - VAS | 12 Months
  Improvement in pain score (Visual Analogue Scale - VAS). Subjects will be asked to rate their pain using a visual analog scale (VAS) from 0-10: 0 = 'no symptoms'; 10 = 'very severe pain'. The amount of improvement in experienced pain is calculated by the following formula: N = [100% × (pre-treatment VAS score-post treatment VAS score)]/pre-treatment VAS score. This result is classified as follows: score 5 = lack of pain or discomfort N=100%; score 4 = marked improvement 75%≤N<100%; scores 3 and 2 = moderate improvement 25%≤N<75%; score 1 = mild improvement 0%<N<25%; score 0 = no improvement N=0.
  The VAS will be monitored both as a daily home-use diary and as a single question at the clinic during the follow-up visits.
Visual Analogue Scale - VAS | 6 Months
  Improvement in pain score (Visual Analogue Scale - VAS). Subjects will be asked to rate their pain using a visual analog scale (VAS) from 0-10: 0 = 'no symptoms'; 10 = 'very severe pain'. The amount of improvement in experienced pain is calculated by the following formula: N = [100% × (pre-treatment VAS score-post treatment VAS score)]/pre-treatment VAS score. This result is classified as follows: score 5 = lack of pain or discomfort N=100%; score 4 = marked improvement 75%≤N<100%; scores 3 and 2 = moderate improvement 25%≤N<75%; score 1 = mild improvement 0%<N<25%; score 0 = no improvement N=0.
  The VAS will be monitored both as a daily home-use diary and as a single question at the clinic during the follow-up visits.
Visual Analogue Scale - VAS | 3 Months
  Improvement in pain score (Visual Analogue Scale - VAS). Subjects will be asked to rate their pain using a visual analog scale (VAS) from 0-10: 0 = 'no symptoms'; 10 = 'very severe pain'. The amount of improvement in experienced pain is calculated by the following formula: N = [100% × (pre-treatment VAS score-post treatment VAS score)]/pre-treatment VAS score. This result is classified as follows: score 5 = lack of pain or discomfort N=100%; score 4 = marked improvement 75%≤N<100%; scores 3 and 2 = moderate improvement 25%≤N<75%; score 1 = mild improvement 0%<N<25%; score 0 = no improvement N=0.
  The VAS will be monitored both as a daily home-use diary and as a single question at the clinic during the follow-up visits.
Oral Lichen Planus (OLP) relapse | 12 Months
  Improvement in OLP relapse rate measured by a decreased need for additional/ repeated treatment with corticosteroid treatment, tacrolimus, or other anti-inflammatory treatment
Use of corticosteroid treatment | 6 Months
  Reduction in the use of corticosteroid treatment according to the anti-inflammatory potency
Graded chronic pain scale (GCPS) questionnaire (authors: Von Korff M et al. 1992) | 12 Months
  Improvement in psychosocial factors assessed by the graded chronic pain scale (GCPS) questionnaire. Grading is based on answering a ten-scale questionnaire from 0, 'no pain' to 10, 'worst possible pain'.
Oral Health Impact Profile (OHIP-14) questionnaire (author: Slade 1997) | 12 Months
  Improvement in psychosocial factors assessed by the oral health impact profile-14 (OHIP-14) questionnaire. The OHIP-14 is a questionnaire that measures people's perception of the social impact of oral disorders on their well-being. Fourteen items of OHIP are divided into seven dimensions: functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability, and handicaps. Grading is based on answering a five-scale questionnaire from 'Never' to 'Very often'.
Generalized anxiety disorder (GAD-7) questionnaire (authors: Spitzer RL et al. 2006) | 12 Months
  Improvement in psychosocial factors assessed by the generalized anxiety disorder (GAD-7) questionnaires. Grading is based on answering a four-scale questionnaire from 0, 'never' to 3, 'almost daily'.
Oral candidosis | 12 Months
  Reduction in number of subjects with oral candidosis during the treatment
Desquamative gingivitis clinical score (DGCS) | 12 Months
  Improvement in OLP measured by the Desquamative Gingivitis Clinical Score (DGCS) by 20 %. The DGCS is a scoring system specifically designed to score the gingival lesions of oral lichen planus. Scoring: 0 = no detectable lesions present; 1 = white lesion; 2 = mild erythema (< 3 mm from gingival margins); 3 = bulla or marked erythema (> 3 mm from gingival margins); 4 = erosion or ulcer

CONTACTS AND LOCATIONS:
Overall Officials: Tommi Pätilä, Docent, Study Director — Chief Medical Officer
Locations (2):
- Finland (2):
  - Tampere University Hospital, Oral and maxillofacial diseases, Tampere, Pirkanmaa
  - Wellbeing services County Pirkanmaa, Health Services, Orthodontics and specialized dental care, Tampere, Pirkanmaa

IPD SHARING:
Plan to Share IPD: No
The IPD will only be administered by the researchers that are listed in the CIP.

REFERENCES:
- See also: Alaijah, F., Morsi, A., Nasher, R. et al. Photobiomodulation therapy in the treatment of periodontal disease: a literature review — https://link.springer.com/article/10.1007/s41547-019-00056-9
- See also: Al-Hashimi I, Schifter M, Lockhart PB, et al., (2007) Oral lichen planus and oral lichenoid lesions: diagnostic and therapeutic considerations — https://pubmed.ncbi.nlm.nih.gov/17261375/
- See also: Akram Z, Javed F, Hosein M, et al., (2018) Photodynamic therapy in the treatment of symptomatic oral lichen planus: A systematic review. — https://pubmed.ncbi.nlm.nih.gov/29223131/
- See also: Arduino PG, Broccoletti R, Sciannameo V, Scully C. (2017) A practical clinical recording system for cases of desquamative gingivitis — https://pubmed.ncbi.nlm.nih.gov/27639053/
- See also: Cheng YS, Gould A, Kurago Z, Fantasia J, Muller S. (2016) Diagnosis of oral lichen planus: a position paper of the American Academy of Oral and Maxillofacial Pathology — https://pubmed.ncbi.nlm.nih.gov/27401683/
- See also: Escudier M, Ahmed N, Shirlaw P, et al., (2007) A scoring system for mucosal disease severity with special reference to oral lichen planus. — https://pubmed.ncbi.nlm.nih.gov/17711534/
- See also: He Y, Deng J, Zhao Y, Tao H et al., (2020) Efficacy evaluation of photodynamic therapy for oral lichen planus: a systematic review and meta-analysis. — https://bmcoralhealth.biomedcentral.com/articles/10.1186/s12903-020-01260-x
- See also: Levine JI. Medications that increase photosensititivity. — http://www.fda.gov/media/75892/download
- See also: Nikinmaa S, Alapulli H, Auvinen P, et al. (2020) Dual-light photodynamic therapy administered daily provides a sustained antibacterial effect on biofilm and prevents Streptococcus mutans adaptation. — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0232775
- See also: Nikinmaa S, Moilanen N, Sorsa T, et al. (2021a). Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. — https://pubmed.ncbi.nlm.nih.gov/34063662/
- See also: Nikinmaa S, Podonyi A, Raivio P, et al. (2021b). Daily Administered Dual-Light Photodynamic Therapy Provides a Sustained Antibacterial Effect on Staphylococcus aureus — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8533018/
- See also: Piboonniyom SO, Treister N, Pitiphat W, Woo SB. (2005) Scoring system for monitoring oral lichenoid lesions: a preliminary study. — https://pubmed.ncbi.nlm.nih.gov/15897856/
- See also: Slade GD (1997) Derivation and validation of a short-form oral health impact profile — https://pubmed.ncbi.nlm.nih.gov/9332805/
- See also: Spitzer RL, Kroenke K, Williams JBW, Löwe B (2006) A brief measure for assessing generalized anxiety disorder: the GAD-7 — https://pubmed.ncbi.nlm.nih.gov/16717171/
- See also: Von Korff M, Ormel J, Keefe FJ, Dworkin SF (1992) Grading the severity of chronic pain — https://pubmed.ncbi.nlm.nih.gov/1408309/
- See also: NICE Guidance IPG615. Low-level laser therapy for preventing or treating oral mucositis caused by radiotherapy or chemotherapy. Interventional procedures guidance [IPG615]. Published: 23 May 2018. — https://www.nice.org.uk/guidance/ipg615